CLINICAL TRIAL: NCT07097259
Title: A Phase 1, Open Label, Randomized, 2-sequence, 2-period, Cross-over, Single Center Study to Assess the Bioequivalence of Follitropin Alfa Solution for Injection in Prefilled Pen (Test) and Follitropin Alfa Powder and Diluent for Solution for Injection in Vial (Reference) in Healthy Downregulated Male Participants
Brief Title: A Study to Assess the Bioequivalence of Follitropin Alfa Solution in Pen and Follitropin Alfa Powder in Vial in Healthy Downregulated Male Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MS700623_0617
Record Dates: First submitted 2025-07-15; First posted 2025-07-31 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Hypogonadism
Keywords: Male Infertility; Follicle Stimulating Hormone
MeSH Terms: conditions — Hypogonadism; Infertility, Male | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Sequence 1 (Experimental): Participants will receive Test follitropin alfa in Period 1 followed by Reference follitropin alfa in Period 2.
  Interventions: Combination Product: Test: Follitropin alfa; Drug: Reference: Follitropin alfa; Drug: Zoladex
- Sequence 2 (Experimental): Participants will receive reference follitropin alfa in Period 1 followed by test follitropin alfa in Period 2.
  Interventions: Combination Product: Test: Follitropin alfa; Drug: Reference: Follitropin alfa; Drug: Zoladex

INTERVENTIONS:
Combination Product: Test: Follitropin alfa — It is a solution for injection in prefilled pen. Participants will receive follitropin alfa on Day 1 in Study Period 1 or Study Period 2. A washout period of at least 23 days will be maintained between period 1 and 2.
Drug: Reference: Follitropin alfa — It is a powder and diluent for solution for injection in multidose vial. Participants will receive follitropin alfa on Day 1 in Study Period 1 or Study Period 2. A washout period of 23 days will be maintained between period 1 and 2.
Drug: Zoladex — It is a auxiliary medicinal product. Participants will receive Zoladex injection on Day -11 in down regulation period, and on Day 17 prior to the start of Period 2.

SUMMARY:
The purpose of this study is to assess the bioequivalence of Test and Reference in healthy downregulated male participants. This is a 2-sequence, 2-period study using the following treatment sequences across Study Periods 1 and 2. At the end of the first Downregulation period (DR1), eligible participants will be randomly assigned to 1 of the 2 treatment sequences:

Sequence 1: Test - Reference Sequence 2: Reference - Test Where, Test = follitropin alfa (solution for injection in prefilled pen), and Reference = follitropin alfa (powder and diluent for solution for injection in vial).

The total duration of the study will be up to approximately 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy, as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring
* Have a normal baseline testosterone level
* Have a body weight of more than equal to 60 kilograms and Body Mass Index within the range 18 to 30 kilograms per meter square
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Any condition, that, in the Investigator's opinion, constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation.
* Participants using the following within 28 days prior to start of study intervention:

  * Drugs or herbal formulations known to increase testosterone levels (e.g. topical testosterone, sildenafil, fluoxymesterone, herbal remedies containing ginseng)
  * Medicinal products known to prolong the QTc interval or medicinal products able to induce torsades de pointes (e.g. antiarrhythmic, antipsychotics, antidepressants, macrolide and quinine antimicrobials, azole antifungals).
* History of clinically relevant cardiovascular events
* History of tumors of the pituitary gland or hypothalamus
* Smokers
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
Baseline Adjusted Area Under the Serum Concentration-Time Curve From Time Zero to Last Quantifiable Sampling Time After Administration (AUC0-t, adj) of Follitropin Alfa | Predose at -45, - 30, -15 minutes, and at 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, (Day 1), 24 and 36 hour (h) (Day 2), 48 h (Day 3), 72 h (Day 4), 96 h (Day 5), 120 h (Day 6), 168 h (Day 8) and 216h (Day 10) after Test/Reference administration
Baseline Adjusted Area Under the Serum Concentration-Time Curve From Time Zero to Infinity (AUC0-inf,adj) of Follitropin Alfa | Predose at -45, - 30, -15 minutes, and at 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, (Day 1), 24 and 36 hour (h) (Day 2), 48 h (Day 3), 72 h (Day 4), 96 h (Day 5), 120 h (Day 6), 168 h (Day 8) and 216h(Day 10) after Test/Reference administration
Baseline Adjusted Maximum Observed Serum Concentration (Cmax,adj) of Follitropin Alfa | Predose at -45, - 30, -15 minutes, and at 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, (Day 1), 24 and 36 hour (h) (Day 2), 48 h (Day 3), 72 h (Day 4), 96 h (Day 5), 120 h (Day 6), 168 h (Day 8) and 216h(Day 10) after Test/Reference administration

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to Day 37
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) by Severity | Up to Day 37
Occurrence of Abnormalities (Grade >=3) in Laboratory Test Values | Up to Day 37
Occurrence of Abnormalities (Grade >=3) in Vital Signs | Up to Day 37
Occurrence of Clinically Significantly Abnormal Electrocardiograms (ECGs) | Up to Day 37
Number of Participants With Local Tolerability/Injection Site Reactions (ISRs) | Up to Day 37
Pharmacokinetic (PK) Plasma Concentrations of Follitropin Alfa | Predose at -45, - 30, -15 minutes, and at 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, (Day 1), 24 and 36 hour (h) (Day 2), 48 h (Day 3), 72 h (Day 4), 96 h (Day 5), 120 h (Day 6), 168 h (Day 8) and 216h(Day 10) after Test/Reference administration
Number of Participants With Positive Anti-Drug Antibody (ADA) of Follitropin Alfa | Predose: Day 1 (Period 1), Day 28 (Period 2), Day 37 (End of Treatment). ADA positive participants followed until end of study(earliest of ADA negative(baseline) or loss to follow-up (upto 40 months)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc.
Locations (1):
- ICON Early Phase Services, LLC_Clinic San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS700623_0617
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html